CLINICAL TRIAL: NCT05823181
Title: Early Versus Late Laparoscopic Exploration of Common Bile Duct After Failure of Extraction of Common Bile Duct Stones by ERCP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Abdelmalak Abd, Principal Investigator, Assiut University
Other Study IDs: CBD stone
Record Dates: First submitted 2023-02-25; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Common Bile Duct Calculi
MeSH Terms: conditions — Gallstones | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early laparoscopic exploration of common bile duct: Early laparoscopic exploration of common bile duct after failure of extraction of common bile duct stones by ERCP
  Interventions: Device: laparoscopy
- Late laparoscopic exploration of common bile duct: late laparoscopic exploration of common bile duct after failure of extraction of common bile duct stones by ERCP
  Interventions: Device: laparoscopy

INTERVENTIONS:
Device: laparoscopy — laparoscopic exploration of common bile duct

SUMMARY:
The goal of this work is to assess the best time to perform LC combined with LCBD exploration and the feasibility and safety of such procedure in patients with combined GBS and CBDS after failure of ERCP extraction of CBD stones .

ELIGIBILITY:
Inclusion Criteria:

1. All patients that presented with calcular obstructive jaundice 2ry to CBD stones.
2. Failed of extraction of common bile duct stone by ERCP.

Exclusion Criteria:

1. patients presented by cholangitis.
2. patients presented by acute pancreatitis.
3. Patients that developed post ERCP pancreatitis ,bleeding , perforation.
4. history of previous biliary surgery rather than cholecystectomy.
5. history of major upper abdominal surgery.
6. pregnant females.
7. patients with liverchirosis, abdominal malignancy , and those unfit for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that presented with calcular obstructive jaundice 2ry to CBD stones and failed of extraction of common bile duct stone by ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
intraoperative complications | Baseline
  1. Assess the operative time in hours
  2. intraoperative blood loss in millilitres
  3. intraoperative organ injury (yes or no)
  4. conversion to open surgery (yes or no)

SECONDARY OUTCOMES:
postoperative complications | Baseline
  1. Postoperative bleeding in millilitres
  2. biliary leakage in millilitres
  3. missed stone (yes or no)
  4. recumbency complications which are monitored for 30 days postoperatively. 5.Overall length of hospital stay and if Intensive Care Unit (ICU) stay needed will also be recorded in days.